CLINICAL TRIAL: NCT03206047
Title: A Randomized Phase 2 Trial of Atezolizumab (MPDL3280A), SGI-110 and CDX-1401 Vaccine in Recurrent Ovarian Cancer
Brief Title: Atezolizumab, Guadecitabine, and CDX-1401 Vaccine in Treating Patients With Recurrent Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01030; NCI-2017-01030 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 285416; 10017 (Other: Roswell Park Cancer Institute EDDOP); 10017 (Other: CTEP); P30CA016056 (NIH)
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Platinum-Resistant Fallopian Tube Carcinoma; Platinum-Resistant Ovarian Carcinoma; Platinum-Resistant Primary Peritoneal Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — atezolizumab; guadecitabine; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort I (atezolizumab) (Experimental): Patients receive atezolizumab IV over 30-60 minutes on days 1 and 15. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Other: Laboratory Biomarker Analysis
- Cohort II (guadecitabine, atezolizumab) (Experimental): Patients receive guadecitabine SC on days 1-5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients also receive atezolizumab IV over 30-60 minutes on days 8 and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Guadecitabine; Other: Laboratory Biomarker Analysis
- Cohort III (guadecitabine, atezolizumab, CDX-1401 vaccine) (Experimental): Patients receive guadecitabine and atezolizumab as in Cohort II. Patients also receive CDX-1401 vaccine IV on day 15 and poly ICLC SC on days 15-16. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Biological: DEC-205/NY-ESO-1 Fusion Protein CDX-1401; Drug: Guadecitabine; Other: Laboratory Biomarker Analysis; Drug: Poly ICLC

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
Biological: DEC-205/NY-ESO-1 Fusion Protein CDX-1401 — Given SC
  Other Names: CDX-1401
  Arms: Cohort III (guadecitabine, atezolizumab, CDX-1401 vaccine)
Drug: Guadecitabine — Given SC
  Other Names: DNMT inhibitor SGI-110; S110; SGI 110; SGI-110; SGI110
  Arms: Cohort II (guadecitabine, atezolizumab); Cohort III (guadecitabine, atezolizumab, CDX-1401 vaccine)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Poly ICLC — Given SC
  Other Names: Hiltonol; Poly I:Poly C with Poly-L-Lysine Stabilizer; poly-ICLC; PolyI:PolyC with Poly-L-Lysine Stabilizer; Polyinosinic-Polycytidylic Acid Stabilized with Polylysine and Carboxymethylcellulose; Polyriboinosinic-Polyribocytidylic Acid-Polylysine Carboxymethylcellulose; Stabilized Polyriboinosinic/Polyribocytidylic Acid
  Arms: Cohort III (guadecitabine, atezolizumab, CDX-1401 vaccine)

SUMMARY:
This randomized phase I/IIb trial studies side effects and best dose of atezolizumab when given together with guadecitabine and CDX-1401 vaccine and to see how well they work in treating patients with ovarian, fallopian tube, or primary peritoneal cancer that has come back. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. CDX-1401 vaccine may enhance the expression of the genes encoding tumor antigens on the surface of tumor cells and enhance the activity of tumor-killing T cells against those tumor cells. Vaccines made from monoclonal antibodies combined with tumor cells may help the body build an effective immune response to kill tumor cells. Giving atezolizumab, guadecitabine, and CDX-1401 vaccine may work better than CDX-1401 alone in treating patients with ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of fixed doses of atezolizumab (MPDL3280A) in combination with guadecitabine (SGI-110). (Phase I) II. To evaluate toxicity of the combination as defined by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. (Phase I) III. To study if SGI-110 improves the benefit of atezolizumab and then if the further addition of the DEC-205/NY-ESO-1 fusion protein CDX-1401 (CDX-1401)/poly ICLC adds further clinical benefit by analyzing progression free survival (PFS), using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. (Phase IIb)

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. (Phase I) II. To determine overall survival (OS), objective response rate (complete and partial responses), clinical benefit rate (response + stable disease), CA-125 reduction (percentage of patients with CA-125 reduction by >= 50%), and duration of response. (Phase IIb) III. To assess the impact of the combination of atezolizumab, SGI-110, and CDX-1401 on anti-tumor immune responses. (Phase IIb) IV. To assess the impact of SGI-110 on NY-ESO-1 expression in tumor tissue. (Phase IIb) V. To assess toxicities associated with the combination cohorts (2 and 3), as there is little human experience with these combinations. (Phase IIb)

EXPLORATORY/TRANSLATIONAL OBJECTIVES:

I. To determine the effectiveness of SGI-110 on enhancing vaccine efficacy by assessing NY ESO 1 specific cellular and humoral immunity.

Ia. Peripheral blood NY ESO 1 specific CD8+ and CD4+ T cells. Ib. Peripheral blood NY ESO 1 specific antibodies. Ic. Peripheral blood unrelated CTA specific antibodies (antigen spreading). Id. Peripheral blood frequency of CD4+CD25+FOXP3+ regulatory T cells. Ie. Examine potential differential effect of NY-ESO-1 expression on PFS. II. To assess the impact on PDL1 expression in tumor tissue. III. Evaluation of therapeutic efficacy on immune cell phenotype. IV. Deoxyribonucleic acid (DNA) methylation and DNA methylome: in pre- and on-treatment peripheral blood, serum (circulating DNA), and tumor biopsies.

V. Pre-and on-treatment density and location of tumor infiltrating CD3+ and CD8+ T cells.

VI. Evaluate the pre- and post-treatment mutational and neo-antigen load and therapeutic efficacy.

VII. Pre- and post-treatment T cell receptor (TCR) repertoire to study the effect of TCR V beta diversity due to combination of PDL1 blockade, epigenetic modification, and vaccination on therapeutic efficacy.

VIII. Gut microbiota at baseline and one on-treatment sample at C4D1 (cycle 4, day 1) or at progression, whichever is earlier to evaluate the role of microbiota on the therapeutic efficacy of the proposed combination therapy.

OUTLINE: This is a phase I, dose-escalation study of guadecitabine followed by a phase IIb study. Patients are randomized to 1 of 3 cohorts.

COHORT I: Patients receive atezolizumab intravenously (IV) over 30-60 minutes on days 1 and 15. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

COHORT II: Patients receive guadecitabine subcutaneously (SC) on days 1-5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients also receive atezolizumab IV over 30-60 minutes on days 8 and 22. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

COHORT III: Patients receive guadecitabine and atezolizumab as in Cohort II. Patients also receive CDX-1401 vaccine IV on day 15 and poly ICLC SC on days 15-16. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 2 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Women with epithelial ovarian, fallopian tube, or primary peritoneal carcinoma with platinum-resistant disease (defined as having relapsed within 6 months of last platinum-containing regimen because we would like to include both primary and secondary resistance); patients are allowed to have had more than 2 prior cytotoxic treatment regimens; all patients should have received standard of care agents, which confer clinical benefit
* Presence of biopsiable disease and patient able to undergo pre-treatment and on-treatment biopsy
* Tissue available from primary and/or recurrent disease to evaluate tumor expression of NY-ESO-1 or PDL1 by immunohistochemistry (IHC) and/or reverse transcriptase-polymerase chain reaction (RT-PCR), and for measurement of DNA methylation
* No requirement for tumor expression of NY-ESO-1
* Life expectancy > 6 months as assessed by study physician
* Because no dosing or adverse event data are currently available on the use of atezolizumab in combination with SGI-110 and CDX-1401 in patients < 18 years of age, children are excluded from this study, but may be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Have been informed of other treatment options
* Have measurable disease outside of biopsy site present per immune related (ir)RECIST criteria; (Rationale: Biopsy may also induce an inflammatory response and bias outcome measurements)
* Patients may have received previous NY ESO 1 vaccine therapy; patients who received bevacizumab or other experimental therapies are eligible for enrollment provided they have discontinued therapy (at least 4 weeks) prior to randomization and recovered from toxicities to less than grade 2
* Leukocytes >= 2,500/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 10 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (however, patients with known Gilbert disease who have serum bilirubin level =< 3 x ULN may be enrolled)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 x ULN (AST and/or ALT =< 3 x ULN for patients with liver involvement)
* Alkaline phosphatase =< 2 x ULN (=< 5 x ULN for patients with documented liver involvement or bone metastases)
* Creatinine clearance >= 30 mL/min/1.73 m^2 by Cockcroft-Gault
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN
* Administration of the drugs used in this study may have an adverse effect on pregnancy and poses a risk to the human fetus, including embryo-lethality; women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 5 months (150 days) after the last dose of study agent; should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Patients who have had chemotherapy or radiotherapy including complementary and alternative medicine treatments (CAMs) within 4 weeks prior to entering the study or those who have not recovered from adverse events (other than alopecia) due to agents administered more than 4 weeks earlier
* Prior treatment with anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents

  * Patients who have received prior treatment with anti-CTLA-4 may be enrolled, provided the following requirements are met:

    * Minimum of 12 weeks from the first dose of anti-CTLA-4 and > 6 weeks from the last dose
    * No history of severe immune-related adverse effects from anti-CTLA-4 (NCI CTCAE grade 3 and 4)
* Treatment with any other investigational agent within 4 weeks prior to cycle 1, day 1
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon [IFN]-alpha or interleukin [IL]-2) within 6 weeks prior to cycle 1, day 1
* Treatment with systemic immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to cycle 1, day 1

  * Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* Patients taking bisphosphonate therapy for symptomatic hypercalcemia; use of bisphosphonate therapy for other reasons (e.g., bone metastasis or osteoporosis) is allowed
* Concomitant systemic treatment with chronic use of anti-histamine or non-steroidal anti-inflammatory drugs and other platelet inhibitory agents and patients on oral anticoagulant (e.g. warfarin); exception: patients on therapeutic anticoagulation therapy such as low-molecular-weight heparin or warfarin at a stable dose level are allowed on study
* Patients with known primary central nervous system (CNS) malignancy or symptomatic CNS metastases are excluded
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* History of allergic reactions attributed to compounds of similar chemical or biological composition to other agents used in this study
* Subjects who have received prior therapy with hypomethylating agents (5-azacytidine, decitabine, SGI-110)
* Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study
* Lack of ability of a patient for immunological and clinical follow-up assessment
* Evidence of current drug or alcohol abuse or psychiatric impairment, which in the investigator's opinion will prevent completion of protocol therapy or follow-up
* Due to unknown effects on the developing fetus or newborn, pregnant or nursing female patients are excluded from this study
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug. (i.e., any significant medical illness or abnormal laboratory finding that would increase the patient's risk by participating in this study)
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA)
* History or risk of autoimmune disease, including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible
  * Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible
  * Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

    * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
    * Rash must cover less than 10% of body surface area (BSA)
    * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%)
    * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan; history of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Patients with active tuberculosis (TB) are excluded
* Severe infections within 4 weeks prior to cycle 1, day 1, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 2 weeks prior to cycle 1, day 1
* Received oral or intravenous (IV) antibiotics within 2 weeks prior to cycle 1, day 1; patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
* Major surgical procedure within 28 days prior to cycle 1, day 1 or anticipation of need for a major surgical procedure during the course of the study
* Administration of a live, attenuated vaccine within 4 weeks before cycle 1, day 1 or anticipation that such a live, attenuated vaccine will be required during the study and up to 5 months after the last dose of atezolizumab

  * Influenza vaccination should be given during influenza season only (approximately October to March); patients must not receive live, attenuated influenza vaccine within 4 weeks prior to cycle 1, day 1 or at any time during the study and until 5 months after the last dose of atezolizumab
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients positive for human immunodeficiency virus (HIV) are NOT excluded from this study, but HIV-positive patients must have:

  * A stable regimen of highly active anti-retroviral therapy (HAART)
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
  * A CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard PCR-based tests
* Patients requiring treatment with a RANKL inhibitor (e.g. denosumab) who cannot discontinue it before treatment with atezolizumab

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AE) (Phase I) | Up to 30 days after last dose
  Will be listed individually per patient according to Common Terminology Criteria for Adverse Events version 5.0, and the number of patients experiencing each AE will be summarized using descriptive statistics.
Progression free survival (PFS) (Phase IIb) | Up to 1 year
  Assessed using standard imaging response (Response Evaluation Criteria in Solid Tumors [RECIST]) criteria. Will be carried forth using a Cox proportional hazards model with a factor for treatment with a stratification factor for disease subtype relative to the determining the form of the likelihood function. The global test statistic will combine from the one-sided tests using Fisher's method for combining p-values. Will also examine potential differential effect of NY-ESO-1 expression on PFS.
  The analysis of expression levels between the three groups will be carried out using analysis-of-variance methods on either the raw values or log transformed values.

SECONDARY OUTCOMES:
Anti-tumor activity (Phase I) | Up to 1 year
  Will observe and record anti-tumor activity.
Overall survival (OS) (Phase IIb) | Up to 1 year
  OS will be measured.
Objective response rate (Phase IIb) | Up to 1 year
  Objective response rate (complete and partial response) will be measured.
Clinical benefit rate (Phase IIb) | Up to 1 year
  Clinical benefit rate (response + stable disease) will be measured.
CA-125 reduction (Phase IIb) | Up to 1 year
  Percentage of patients with CA-125 reduction by >= 50% will be measured. Continuous endpoints will be analyzed using the Kruskal-Wallis rank-sum test.
Duration of response (Phase IIb) | Up to 1 year
  Duration of response will be measured.
Anti-tumor immune responses (Phase IIb) | Up to 1 year
  The impact of the combination of atezolizumab, guadecitabine, and CDX-1401 on anti-tumor immune responses will be measured.
Epigenetic modification of immune gene signatures, NY-ESO-1, other CTAs, and PDL1 in the tumor microenvironment (Phase IIb) | Up to 1 year
  Epigenetic modification of immune gene signatures, NY-ESO-1, other CTAs, and PDL1 in the tumor microenvironment will be assessed.
Incidence of adverse events with the combination cohorts (2 and 3) (Phase IIb) | Up to 30 days after last dose
  According to Common Terminology Criteria for Adverse Events version 5.0.

OTHER OUTCOMES:
NY-ESO-1-specific immune responses | Up to 1 year
  Will be assessed by enzyme-linked immunosorbent spot assay and fluorescence activated cell sorting on NY-ESO-1-specific T cells.
PDL1 expression in tumor tissue | Up to 1 year
  Will be assessed by immunohistochemistry.
AIM gene signatures | Up to 1 year
  Will be assessed by Nanostring immune profiling panel.
Immune cell phenotype | Up to 1 year
  Will be assessed by fluorescence activated cell sorting.
Neo-antigen and mutational antigen | Up to 1 year
  Will be assessed by whole exome sequencing and ribonucleic acid (RNA) sequencing.
T cell receptor (TCR) repertoire | Up to 1 year
  Will be assessed by TCR sequencing for V-beta.
Microbiome | Up to 1 year
  Will be assessed by microbiome sequencing and bacterial 16s RNA expression.

CONTACTS AND LOCATIONS:
Overall Officials: Kunle Odunsi, Principal Investigator — Roswell Park Cancer Institute EDDOP
Locations (17):
- United States (17):
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah